CLINICAL TRIAL: NCT00027378
Title: Pharmacological Intervention Project (Fluoxetine)
Acronym: FIDAA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jack Cornelius, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIAAACOR13370; R01AA015173 (NIH); R01AA013370 (NIH); AA-13370
Record Dates: First submitted 2001-12-04; First posted 2001-12-05 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-06

CONDITIONS: Alcoholism; Depression
Keywords: fluoxetine,; adolescents,; alcohol dependence,; major depression; Alcoholism
MeSH Terms: conditions — Alcoholism; Depression; Depressive Disorder, Major | interventions — Fluoxetine; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): fluoxetine plus Treatment As Usual (TAU)
  Interventions: Drug: fluoxetine (Prozac)
- 2 (Placebo Comparator): placebo plus Treatment As Usual (TAU)
  Interventions: Drug: Placebo plus Treatment As Usual

INTERVENTIONS:
Drug: fluoxetine (Prozac) — fluoxetine plus Treatment As Usual (TAU); 12 weeks acute phase; plus 9 month naturalistic follow up
  Arms: 1
Drug: Placebo plus Treatment As Usual — placebo plus Treatment as Usual; 12 weeks acute phase; plus 9 month naturalistic follow up
  Arms: 2

SUMMARY:
This is a large scale study involving fluoxetine (Prozac) versus a placebo in the treatment of adolescents with alcohol use disorder (AUD) and major depression (MDD). All individuals will receive treatment for 12 weeks with a followup phase lasting 9 months.

DETAILED DESCRIPTION:
Recently, the first large-scale double-blind, placebo-controlled study of a selective serotonin reuptake inhibitor (SSRI) antidepressant in depressed adolescents was completed (Emslie et al., 1997) That study demonstrated efficacy for fluoxetine in non-AUD adolescents with major depressive disorder (MDD). Our own research group recently completed a first double-blind, placebo-controlled study of fluoxetine in adults with comorbid MDD and alcohol dependence (Cornelius et al., 1997). That study demonstrated efficacy for fluoxetine in decreasing both the depressive symptoms and the alcohol use of adult depressed alcoholics. Our own research group also recently completed a pilot study involving open label fluoxetine in adolescents with comorbid AUD and MDD. That pilot study demonstrated within-group efficacy for fluoxetine for decreasing both the drinking and the depressive symptoms of that population, and suggested that fluoxetine is a safe medication in this population (Cornelius, et al., In Press). However, to date, no double-blind, placebo-controlled study of any selective serotonin re-uptake inhibitors (SSRI) medication has been conducted in adolescents with a comorbid AUD and MDD. In this proposed study, a first large scale prospective double-blind, placebo-controlled study will be undertaken involving the SSRI medication fluoxetine versus placebo in the treatment of adolescents with an alcohol use disorder and major depression (AUD/MDD).

The goals of the study include the following: 1) to compare the efficacy of the SSRI medication fluoxetine plus Treatment As Usual (TAU) to placebo plus TAU for the alcohol use and the depressive symptoms of an adolescent sample (ages 15 to 18) of subjects with comorbid diagnoses of an AUD and MDD; 2) to assess specific predictors of medication response in that study; and to perform a preliminary evaluation of the longer-term efficacy of fluoxetine in these patients, in a 9-month naturalistic follow-up period beyond the 3 month acute phase study. We hypothesize that fluoxetine plus TAU will demonstrate efficacy for decreasing both the drinking and the depressive symptoms of this population.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol use disorder and major depressive disorder.

Exclusion Criteria:

* Meets criteria for bipolar disorder, schizoaffective disorder, or schizophrenia.
* Hyper- or hypothyroidism, significant cardiac, neurologic, or renal impairment, and those with significant liver disease.
* Receiving antipsychotic or antidepressant medication in the month prior to entering the study.
* Use of any illicit substance abuse or dependence other than cannabis abuse (and alcohol abuse).
* History of intravenous drug use.
* Pregnancy, inability or unwillingness to use contraceptive methods.
* Inability to read or understand study forms
* Less than 15 years of age or over 18 years of age will be excluded.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2001-07; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Cornelius, M.D., Principal Investigator — Western Psychiatric Institute and Clinic Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Cornelius JR, Bukstein OG, Wood DS, Kirisci L, Douaihy A, Clark DB. Double-blind placebo-controlled trial of fluoxetine in adolescents with comorbid major depression and an alcohol use disorder. Addict Behav. 2009 Oct;34(10):905-9. doi: 10.1016/j.addbeh.2009.03.008. Epub 2009 Mar 12. PMID 19321268

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Western Psychiatric Institute and Clinic (WPIC) of the University of Pittsburgh Medical Center (UPMC). Subjects were recruited for participation in the treatment study through referrals from any of the WPIC treatment programs and by responding to newspaper, radio and bus advertisements.
Pre-assignment Details: Exclusion: bipolar disorder, schizoaffective disorder, schizophrenia, hyper-or hypothyroidism, cardiac, neurological, renal impairment, significant liver disease, received antipsychotic or antidepressant medication, substance abuse or dependence, intravenous drug use, pregnancy, inability or unwillingness to use contraceptive methods, illiteracy.
Groups:
- Fluoxetine Plus Treatment As Usual (TAU): Subjects were treated with the medication fluoxetine (15 mg to 30 mg) plus Treatment as Usual (TAU), which included Cognitive Behavioral Therapy and Motivational Enhancement Therapy (CBT/MET) psychotherapy.
- Placebo Plus Treatment as Usual (TAU): Subjects were treated with placbo plus Treatment as Usual (TAU), which included Cognitive Behavioral Therapy and Motivational Enhancement Therapy (CBT/MET) psychotherapy.
Period: Overall Study
Arm/Group | Fluoxetine Plus Treatment As Usual (TAU) | Placebo Plus Treatment as Usual (TAU)
Started | 24 | 26
Completed | 24 | 23
Not Completed | 0 | 3
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine Plus Treatment As Usual (TAU) | Placebo Plus Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 22 | 25 | 47
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 19.5 (.94) | 19.4 (.91) | 19.4 (.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use Behaviors
Description: Alcohol use behaviors measured by drinks per week.
Time Frame: Average number of drinks as recorded on the Timeline Follow-Back (subject-reported) measure daily over the 12-week acute phase.
Population: Participants were randomized to either fluoxetine-treated or placebo.
Measure: Mean (Standard Deviation); unit: standard drink (14 gr. alcohol)
Arm/Group | Fluoxetine Plus Treatment As Usual (TAU) | Placebo Plus Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 26
standard drink (14 gr. alcohol) | 1.56 (1.44) | 1.73 (1.61)
Statistical Analysis 1: Comparison: Fluoxetine Plus Treatment As Usual (TAU) vs Placebo Plus Treatment as Usual (TAU); Repeated measures ANOVA; Test type: Superiority or Other; p = .05, ANOVA; repeated measures; Mean Difference (Final Values) = 0.39, Standard Deviation 0.702

2. Primary Outcome: Depressive Symptoms
Description: Beck Depression Inventory (BDI) Scores measured at Weeks 1-4, 6, 8, 10, 12. The BDI is a subject reported measure that has a minimum score of 0 and a maximum score of 63. A better outcome would consist of values near the minimum end of the scale (0) and a worse outcome would consist of values near the maximum end of the scale (63).
Time Frame: Average score as measured by participant's report on the Beck Depression Inventory (BDI).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine Plus Treatment As Usual (TAU) | Placebo Plus Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 26
units on a scale | 6.79 (7.49) | 10.46 (10.80)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked during the 12-week acute treatment phase.
Arm/Group | Fluoxetine Plus Treatment As Usual (TAU) | Placebo Plus Treatment as Usual (TAU)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

LIMITATIONS AND CAVEATS:
Limited sample size; efficacy of CBT/MET Therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No